CLINICAL TRIAL: NCT03245229
Title: A Single-center, Open-label, One-sequence, Two-treatment Study to Investigate the Effect of ACT-132577 at Steady State on the Pharmacokinetics of Rosuvastatin in Healthy Male Subjects
Brief Title: A Study in Healthy Male Subjects to Investigate Whether Administration of ACT-132577 Can Affect Rosuvastatin's Fate in the Body (Amount and Time of Presence in the Blood)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC-080-106
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — aprocitentan; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): In the morning of Day 1, a single dose of 10 mg rosuvastatin will be administered in the fasted state followed by an observation period of 96 h
  Interventions: Drug: Rosuvastatin
- Treatment B1 (Experimental): 25 mg ACT-132577 will be administered o.d. from Day 5 to Day 12
  Interventions: Drug: Aprocitentan
- Treatment B2 (Experimental): In the morning of Day 13, a single dose of 10 mg rosuvastatin will be administered in the fasted state, concomitantly with 25 mg ACT-132577, followed by an observation period of 120 h.
  Doses of 25 mg ACT-132577 will be administered o.d. from Day 14 to Day 17.
  Interventions: Drug: Aprocitentan; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Aprocitentan — Capsule for oral administration
  Other Names: ACT-132577
  Arms: Treatment B1; Treatment B2
Drug: Rosuvastatin — Tablet for oral administration
  Arms: Treatment A; Treatment B2

SUMMARY:
The primary purpose of this study is to investigate the effect of Aprocitentan (ACT-132577) at steady state on the pharmacokinetics of single-dose rosuvastatin in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study mandated procedure;
* Healthy male subjects aged 18 to 45 years (inclusive) at screening;
* Body mass index of 18.0 to 28.0 kg/m2 (inclusive) at screening;
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests;
* Hemoglobin ≥ 135 g/L at screening.

Exclusion Criteria:

* Known allergic reactions or hypersensitivity to ACT-132577, rosuvastatin, any drug of the same classes, or any of their excipients;
* Any contraindication for rosuvastatin treatment;
* History or clinical evidence of myopathy;
* Asian or Indian-Asian ethnicity;
* Known hypersensitivity or allergy to natural rubber latex;
* Previous exposure to ACT-132577;
* Treatment with rosuvastatin within 3 months prior to screening;
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of rosuvastatin | Up to Day 29
  Cmax of rosuvastatin will be derived by non-compartmental analysis of the plasma concentration-time profiles
Time to reach Cmax (tmax) of rosuvastatin | Up to Day 29
  tmax of rosuvastatin will be derived by non-compartmental analysis of the plasma concentration-time profiles
Terminal half-life (t1/2) of rosuvastatin | Up to Day 29
  t1/2 of rosuvastatin will be derived by non-compartmental analysis of the plasma concentration-time profiles
Area under the plasma concentration-time curves during a dosing interval [AUC(0-t)] of rosuvastatin | Up to Day 29
  AUC(0-t) of rosuvastatin will be derived by non-compartmental analysis of the plasma concentration-time profiles
Area under the plasma concentration-time curves from time 0 to inf [AUC(0-inf)] of rosuvastatin | Up to Day 29
  AUC(0-inf) of rosuvastatin will be derived by non-compartmental analysis of the plasma concentration-time profile
Trough (pre-dose) plasma concentrations (Ctrough) of ACT-132577 | Up to Day 29
  Ctrough of ACT-132577 will be derived by non-compartmental analysis of the plasma concentration-time profile

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to Day 29
  Treatment emergent adverse events and treatment emergent serious adverse events will be evaluated throughout the study
Changes from baseline in electrocardiogram (ECG) variables | Up to Day 29
  ECG variables are to be recorded at rest using a standard 12-lead ECG
Changes from baseline in blood pressure | Up to Day 29
  Blood pressure (mmHg) measured using an automatic oscillometric device
Changes from baseline in pulse rate | Up to Day 29
  Pulse rate (bpm) measured using an automatic oscillometric device

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Cepha s.r.o, Pilsen, Czechia